CLINICAL TRIAL: NCT01396239
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Efficacy, Safety, Tolerability and Pharmacokinetics Study of AVI-4658(Eteplirsen),in the Treatment of Ambulant Subjects With Duchenne Muscular Dystrophy
Brief Title: Efficacy Study of AVI-4658 to Induce Dystrophin Expression in Selected Duchenne Muscular Dystrophy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4658-us-201; 07-2484 (Other: Office of Orphan Drug Development)
Record Dates: First submitted 2011-07-08; First posted 2011-07-18 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVI-4658 (Eteplirsen) (Experimental): 1. 50 mg/kg eteplirsen for 28 weeks
  2. 30 mg/kg eteplirsen for 28 weeks
  Interventions: Drug: AVI-4658 (Eteplirsen)
- Placebo / Delayed Treatment (Placebo Comparator): 3a. Placebo 50 mg/kg phosphate buffered saline solution identical in appearance to eteplirsen for 24 weeks followed by 50 mg/kg of eteplirsen for 4 weeks.
  3b. Placebo 30 mg/kg phosphate buffered saline solution identical in appearance to eteplirsen for 24 weeks followed by 30 mg/kg of eteplirsen for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AVI-4658 (Eteplirsen) — Treatment group 1 (n=4): 50.0 mg/kg eteplirsen once weekly x 24 weeks via a 60-minute i.v. infusion Treatment group 2 (n=4): 30.0 mg/kg eteplirsen once weekly x 24 weeks via a 60-minute i.v. infusion Treatment group 3 (n=4): matching placebo once weekly x 24 weeks via a 60-minute i.v. infusion; treatment group 3a will match two placebo subjects to 50.0 mg/kg eteplirsen; treatment group 3b will match two placebo subjects to 30.0 mg/kg eteplirsen
  Other Names: Eteplirsen- Phosphorodiamidate Morphilino Oligomer
  Arms: AVI-4658 (Eteplirsen)
Other: Placebo — sterile, isotonic, clear, colorless phosphate buffered saline solution of eteplirsen at a concentration of 100 mg/mL in single-use vials containing a nominal volume of 1.0 mL without preservatives.
  Other Names: Phosphate buffered saline
  Arms: Placebo / Delayed Treatment

SUMMARY:
This study is designed to assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of AVI-4658 (eteplirsen) in both 50.0 mg/kg and 30.0 mg/kg doses administered over 24 weeks in subjects diagnosed with Duchenne muscular dystrophy (DMD).

DETAILED DESCRIPTION:
For details regarding the roll-over extension study 4658-us-202, please refer to NCT01540409.

ELIGIBILITY:
Major Inclusion and Exclusion Criteria:

Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for this study.

* Be a male with DMD and have an out-of-frame deletion(s) that may be corrected by skipping exon 51 [e.g., deletions of exons 45-50, 47-50, 48-50, 49-50, 50, 52, 52-63], as confirmed in a Clinical Laboratory Improvement Act-accredited laboratory by any of the peer-reviewed and published methodology that evaluates all exons (including, but not limited to, multiplex ligation-dependent probe, comparative genomic hybridization, and single condition amplification/internal primer analysis).
* Be between the ages of 7 and 13 years, inclusive.
* Have stable cardiac function and stable pulmonary function (forced vital capacity [FVC] ≥50% of predicted and not require supplemental oxygen) that, in the Investigator's opinion, is unlikely to decompensate over the duration of the study.
* Be receiving treatment with oral corticosteroids and have been on a stable dose for at least 24 weeks before study entry. Subjects may be allowed to take other (non-RNA antisense or gene therapy) medication (including angiotensin-converting enzyme [ACE] inhibitors, β blockers, losartan potassium, and coenzyme Q) as long as they have been on a stable dose of the medication for 24 weeks before the screening visit (Visit 1) and the dose will remain constant throughout the study.
* Have intact right and left biceps muscles or an alternative upper arm muscle group.
* Achieve an average distance within 200m and 400m ±10% (i.e. within 180m and 440m) while walking independently over six minutes.
* Have a left ventricular ejection fraction (LVEF) of >40% based on the ECHO that is obtained at the screening visit (Visit 1). A subject who has abnormal ECHO findings but who has an LVEF of >40% may be enrolled in the study at the Investigator's discretion; however, the subject must have been receiving stable doses of ACE inhibitors or β blockers for at least 24 weeks before study entry.
* Have a parent(s) or legal guardian(s) who is able to understand and comply with the all of the study procedure requirements.
* Be willing to provide informed assent and have a parent(s) or legal guardian(s) who is willing to provide written informed consent for the subject to participate in the study.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from this study.

* Use of any pharmacologic treatment, other than corticosteroids, that might have an effect on muscle strength or function within 12 weeks before study entry (e.g., growth hormone, anabolic steroids).
* Previous treatment with the experimental agents eteplirsen, BMN-195, or PRO051.
* Previous treatment with any other experimental agents or participation in any other DMD interventional clinical study within 12 weeks before entry into this study; including use of the shock training system or "STS," or planned use during this study.
* Surgery within 3 months before study entry or planned surgery at any time during this study.
* Presence of other clinically significant illness at the time of study entry, including significant renal dysfunction (as measured by urinary cystatin C, KIM-1, or urinary total protein), or average heart rate during screening Holter monitoring in excess of 110 bpm (unless subsequently treated and confirmed controlled and stable on a β-blocker) or QTc >450 ms.
* Use of any aminoglycoside antibiotic within 12 weeks before the screening visit (Visit 1) or need for use of an aminoglycoside antibiotic during the study (unless discussed and agreed with the Principal Investigator and medical monitor).
* Prior or ongoing medical condition that, in the Investigator's opinion, could adversely affect the safety of the subject or that makes it unlikely that the course of treatment or follow-up would be completed or could impair the assessment of study results.

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Mendell JR, Goemans N, Lowes LP, Alfano LN, Berry K, Shao J, Kaye EM, Mercuri E; Eteplirsen Study Group and Telethon Foundation DMD Italian Network. Longitudinal effect of eteplirsen versus historical control on ambulation in Duchenne muscular dystrophy. Ann Neurol. 2016 Feb;79(2):257-71. doi: 10.1002/ana.24555. Epub 2016 Jan 8. PMID 26573217
- [Derived] Mendell JR, Rodino-Klapac LR, Sahenk Z, Roush K, Bird L, Lowes LP, Alfano L, Gomez AM, Lewis S, Kota J, Malik V, Shontz K, Walker CM, Flanigan KM, Corridore M, Kean JR, Allen HD, Shilling C, Melia KR, Sazani P, Saoud JB, Kaye EM; Eteplirsen Study Group. Eteplirsen for the treatment of Duchenne muscular dystrophy. Ann Neurol. 2013 Nov;74(5):637-47. doi: 10.1002/ana.23982. Epub 2013 Sep 10. PMID 23907995
- See also: Mendell, 2013, Annals of Neurology — http://www.ncbi.nlm.nih.gov/pubmed/?term=23907995
- See also: Mendell, 2016, Annals of Neurology — http://www.ncbi.nlm.nih.gov/pubmed/?term=26573217
- See also: Kinane, 2018, Journal of Neuromuscular Diseases — http://www.ncbi.nlm.nih.gov/pubmed/?term=Kinane+eteplirsen
- See also: Charleston, 2018, Neurology — http://www.ncbi.nlm.nih.gov/pubmed/29752304
- See also: Cirak, Lancet, 2001 — http://www.ncbi.nlm.nih.gov/pubmed/21784508

RESULTS

PARTICIPANT FLOW:
Groups:
- AVI-4658 (Eteplirsen) 50 mg/kg: 50 mg/kg eteplirsen for 24 weeks
- Placebo - Week 12 Biopsy: Placebo for 24 Weeks with muscle Biopsy at Week 12
- AVI-4658 (Eteplirsen) 30 mg/kg: 30 mg/kg eteplirsen for 24 weeks
- Placebo - Week 24 Biopsy: Placebo for 24 weeks with muscle biopsy at Week 24
Period: Overall Study
Arm/Group | AVI-4658 (Eteplirsen) 50 mg/kg | Placebo - Week 12 Biopsy | AVI-4658 (Eteplirsen) 30 mg/kg | Placebo - Week 24 Biopsy
Started | 4 | 2 | 4 | 2
Completed | 4 | 2 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo: phosphate buffered saline solution identical in appearance to eteplirsen for 24 weeks
- Total: Total of all reporting groups
Arm/Group | AVI-4658 (Eteplirsen) 30 mg/kg | AVI-4658 (Eteplirsen) 50 mg/kg | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 4 | 12
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (0.50) | 8.5 (1.29) | 8.5 (1.73) | 8.8 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number (%) of Dystrophin Positive Fibers
Description: The primary efficacy endpoint will be based on the pre-treatment and post-treatment change in the number (%) of dystrophin positive fibers as measured in the muscle biopsy tissue on immunohistochemistry (IHC).
Time Frame: After 12 weeks for 4 patients who received 50 mg/kg and 2 patients who received placebo. After 24 weeks for 4 patients who received 30 mg/kg and 2 patients who received placebo.
Population: The sample size for the study was selected based on Proof of Principal approach.
Measure: Least Squares Mean (Full Range); unit: percentage of dystrophin Pos. fibers
Groups:
- AVI-4658 (Eteplirsen) 30 mg/kg: 30 mg/kg eteplirsen - Biopsied after 24 weeks of dosing
- Placebo - Week 24 Biopsy: Placebo: Biopsied after 24 weeks of dosing
- AVI-4658 (Eteplirsen) 50 mg/kg: 50 mg/kg eteplirsen - Biopsied after 12 weeks of dosing
- Placebo - Week 12 Biopsy: Placebo - Biopsied after 12 weeks of dosing
Arm/Group | AVI-4658 (Eteplirsen) 30 mg/kg | Placebo - Week 24 Biopsy | AVI-4658 (Eteplirsen) 50 mg/kg | Placebo - Week 12 Biopsy
Number analyzed (Participants) | 4 | 2 | 4 | 2
percentage of dystrophin Pos. fibers | 23 [15.9 to 29.0] | -7.48 [-8.5 to -6.5] | 0.79 [-9.3 to 7.4] | -0.63 [-5.8 to 4.5]

2. Secondary Outcome: Change From Baseline: 6 Minute Walk Test (6MWT) - Intent to Treat Population (ITT)
Description: A key secondary efficacy endpoint will be based on the pre-treatment and post-treatment Change from baseline: 6 Minute Walk Test (6MWT) - Intent to Treat population (ITT)
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: Meters
Groups:
- 30 mg/kg Eteplirsen: 30 mg/kg eteplirsen for 24 weeks
- 50 mg/kg Eteplirsen: 50 mg/kg eteplirsen for 24 weeks
- Placebo: Placebo for 24 weeks
Arm/Group | 30 mg/kg Eteplirsen | 50 mg/kg Eteplirsen | Placebo
Number analyzed (Participants) | 4 | 4 | 4
Meters | -134.8 (72.36) | -2.3 (14.95) | -17.3 (14.03)

3. Secondary Outcome: Change From Baseline: 6 Minute Walk Test (6MWT) - Modified Intent to Treat Population (mITT)
Description: A key secondary efficacy endpoint will be based on the pre-treatment and post-treatment of the 6-MWT distance. Change from baseline: 6 Minute Walk Test (6MWT) - modified Intent-to-Treat population (mITT).
Time Frame: 24 weeks
Population: The mITT population excludes 2 patients in the 30mg/kg arm who showed rapid disease progression within weeks of enrollment, and were unable to complete assessments that required ambulation at or beyond Week 24.
Measure: Mean (Standard Error); unit: Meters
Groups:
- 30mg/kg Eteplirsen: 30mg/kg eteplirsen for 24 weeks
- 50mg/kg Eteplirsen: 50mg/kg eteplirsen for 24 weeks
Arm/Group | 30mg/kg Eteplirsen | 50mg/kg Eteplirsen | Placebo
Number analyzed (Participants) | 2 | 4 | 4
Meters | -12.5 (1.50) | -2.3 (14.95) | -17.3 (14.03)

4. Post Hoc Outcome: Adverse Events >30%
Description: Adverse events that occurred in >30% of the overall patient population across treatment arms.
Time Frame: 24 Weeks
Measure: Number; unit: Number of patients
Groups:
- AVI-4658 (Eteplirsen) - 30mg/kg: 30 mg/kg eteplirsen for 24 weeks
- AVI-4658 (Eteplirsen) - 50mg/kg: 50 mg/kg eteplirsen for 24 weeks
- Placebo: Placebo for 24 weeks - Phosphate buffered saline solution identical in appearance to eteplirsen
Arm/Group | AVI-4658 (Eteplirsen) - 30mg/kg | AVI-4658 (Eteplirsen) - 50mg/kg | Placebo
Number analyzed (Participants) | 4 | 4 | 4
Number of patients
  Procedural Pain | 1 | 3 | 3
  Oropharyngeal Pain | 3 | 0 | 3
  Hypokalemia (a known side effect of steroids) | 2 | 2 | 2
  Cough | 1 | 1 | 2
  Extremity Pain | 0 | 1 | 3

5. Post Hoc Outcome: Frequency of AEs Related to Eteplirsen
Description: Frequency of AEs that the study physician considered to be any of the following: Related; Possibly related; or Probably related to eteplirsen.
Time Frame: 24 Weeks
Measure: Number; unit: Number of patients
Arm/Group | AVI-4658 (Eteplirsen) - 30mg/kg | AVI-4658 (Eteplirsen) - 50mg/kg | Placebo
Number analyzed (Participants) | 4 | 4 | 4
Number of patients
  Intermittent Nausea (mild) | 0 | 0 | 1
  Other AEs related to eteplirsen | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | AVI-4658 (Eteplirsen) - 30mg/kg | AVI-4658 (Eteplirsen) - 50mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVI-4658 (Eteplirsen) - 30mg/kg (N=4) | AVI-4658 (Eteplirsen) - 50mg/kg (N=4) | Placebo (N=4)
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Balance Disorder (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Haematoma (Vascular disorders) | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Injection Site Pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Enterobiasis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Uticaria thermal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the small number of study participants, a single adverse event (AE) in 1 patient exceeds the reporting threshold of 5%. Refer to the "Post-Hoc Outcome Measures" #4 and #5 for a summary of frequent and related AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Non Disclosure Agreement provides that the PI, Dr. Jerry Mendell, cannot disclose any "results of the discussions or evaluation" without our consent, and that the "proprietary information shall not be evaluated by any laboratory or clinical testing or experimentation conducted" without our consent.